CLINICAL TRIAL: NCT00739700
Title: Accuracy and Precision of Oscillometric Blood Pressure Monitoring in the Arm, Calf and Thighs of Medical ICU Patients When Compared to Invasive Arterial Blood Pressure Monitoring
Brief Title: Non-invasive Blood Pressure (BP) Monitoring Compared to A-Line BP Monitoring
Acronym: NIBP vs IABP
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00001777
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-01

CONDITIONS: Blood Pressure
Keywords: hemodynamics; blood pressure; blood pressure monitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: There is only one cohort of subjects, the critically ill. The NIBP will be correlated with the IABP in each subject.

SUMMARY:
Blood pressure cuffs (NIBP) are slowly replacing intra-arterial (IABP) measurement as the standard of care in the medical intensive care unit. There is little data to support this clinical normalization of deviance. This study aims to correlate NIBP with IABP.

DETAILED DESCRIPTION:
It has become standard practice in inpatient and intensive care settings to monitor systolic, diastolic and mean arterial blood pressure by oscillometric technique. Several studies have confirmed the accuracy and precision of the oscillometric technique in ambulatory patients at both the level of the brachial and radial arteries. Multiple clinical research studies have demonstrated that when blood pressures (systolic, diastolic and mean arterial pressures) determined by non-invasive blood pressure monitors (NIBP) from various manufacturers are compared to direct invasive arterial pressure monitors, the two values are on average within 5 mm Hg of each other. There is limited data in critically ill patients. To date, there are no studies evaluating the accuracy or precision of these devices in intensive care patients for alternative sites (calf, thigh). In addition, there are no large clinical studies evaluating oscillometric NIBP monitoring in a complex medical intensive care population with varying hemodynamics. The goal of this study is to validate the oscillometric technique in measurement of blood pressure in the calf and thigh regions when compared to a gold standard. We may also be able to evaluate more specifically which situations for our patient population the blood pressure will be accurately portrayed as compared with the arterial pressure tracing. It has possible clinical value in either validating non-invasive blood pressure monitoring and eliminating/decreasing the need for invasive arterial blood pressure monitoring. Our hypothesis is that NIBP in the medical intensive care patients is highly variable and not a reliable means of arterial blood pressure monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Arterial blood pressure line

Exclusion Criteria:

* Lack of arms and legs for cuff pressures
* Medical or surgical indication that might prevent use of blood pressure cuffs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical Intensive Care Unit patients with intra-arterial blood pressure catheters will be enrolled. Blood pressure cuff measurements will be made in both arms and both legs.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Correlation between NIBP and IABP. NIBP is measured in both upper arms, both wrists, both thighs, and both ankles. | All NIBP's are measured within 10 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Arjun B Chatterjee, MD, MS, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
A requestor must have local IRB approval and funding to support a request of this data. It will be provided de-identified and shared authorship is required.

REFERENCES:
- [Background] Bur A, Hirschl MM, Herkner H, Oschatz E, Kofler J, Woisetschlager C, Laggner AN. Accuracy of oscillometric blood pressure measurement according to the relation between cuff size and upper-arm circumference in critically ill patients. Crit Care Med. 2000 Feb;28(2):371-6. doi: 10.1097/00003246-200002000-00014. PMID 10708169
- [Background] Bur A, Herkner H, Vlcek M, Woisetschlager C, Derhaschnig U, Delle Karth G, Laggner AN, Hirschl MM. Factors influencing the accuracy of oscillometric blood pressure measurement in critically ill patients. Crit Care Med. 2003 Mar;31(3):793-9. doi: 10.1097/01.CCM.0000053650.12025.1A. PMID 12626986
- [Background] Davis JW, Davis IC, Bennink LD, Bilello JF, Kaups KL, Parks SN. Are automated blood pressure measurements accurate in trauma patients? J Trauma. 2003 Nov;55(5):860-3. doi: 10.1097/01.TA.0000092686.91877.DE. PMID 14608157
- [Background] Chatterjee A, DePriest K, Blair R, Bowton D, Chin R. Results of a survey of blood pressure monitoring by intensivists in critically ill patients: a preliminary study. Crit Care Med. 2010 Dec;38(12):2335-8. doi: 10.1097/CCM.0b013e3181fa057f. PMID 20890190
- [Background] DePriest KL, Cauthen CG, Perry CD, Blair RA, Chatterjee A, Bowton D, Chin R. Do oscillatory blood pressure measurements in upper and lower extremities correlate in patients in the intensive care unit? Chest. 2008; 134(4_Meeting Abstracts): 119001.